CLINICAL TRIAL: NCT04909190
Title: A Randomized Trial of an Increased Saline Flush Protocol to Reduce the Amount of Residual Air Inside a Stentgraft Delivery System
Brief Title: Saline Flush to Reduce the Amount of Residual Air Inside a Stentgraft Delivery System
Acronym: SAFRANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Csaba Csobay-Novák MD PhD, Chief radiologist, Noninvasive Imaging, Semmelweis University Heart and Vascular Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SF2021
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Aortic Aneurysm; Aortic Aneurysm, Thoracic; Aortic Diseases; Aortic Arch Aneurysm; Stroke
Keywords: endovascular; evar; tevar; stentgraft; de-airing
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Thoracic; Aortic Diseases; Aneurysm, Aortic Arch; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1xIFU (No Intervention): Subjects in this arm are randomized to have a saline flush volume according to the IFU of the used device.
- 4xIFU (Experimental): Subjects in this arm are randomized to have a saline flush volume of 4x of what is stated in the IFU of the used device.
  Interventions: Procedure: Increased saline flush volume

INTERVENTIONS:
Procedure: Increased saline flush volume — Additional flushing of the stentgraft delivery system.
  Arms: 4xIFU

SUMMARY:
Non-randomized studies have shown that de-airing of the delivery system with an increased volume of saline may be associated to a decrease in periprocedural stroke during thoracic endovascular aortic repair. This study is designed to provide evidence that 4xIFU-dose volume of saline flush vs. standard IFU-dose saline flush is associated to a decrease in the amount of intra-sac air detected on the first follow-up imaging after EVAR.

ELIGIBILITY:
Inclusion Criteria:

* endovascular aortic repair of an abdominal aortic aneurysm using either of these devices: Terumo/Bolton Treo, Terumo Anaconda, Cook Zenith Alpha Abdominal

Exclusion Criteria:

* concomitant use of an iliac bifurcation device due to insufficient common iliac landing zone on either side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Air volume | within 7 days after index procedure
  Total volume of air inside the aneurysm sac on discharge CT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Csobay-Novák, MD PhD, Study Director — Dept. of Interventional Radiology, Heart and Vascular Center, Semmelweis University
Locations (1):
- Heart and Vascular Center, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szentivanyi A, Borzsak S, Vecsey-Nagy M, Suvegh A, Huttl A, Fontanini DM, Szeberin Z, Csobay-Novak C. The impact of increasing saline flush volume to reduce the amount of residual air in the delivery system of aortic prostheses-a randomized controlled trial. Front Cardiovasc Med. 2024 Mar 22;11:1335903. doi: 10.3389/fcvm.2024.1335903. eCollection 2024. PMID 38586170